CLINICAL TRIAL: NCT07146698
Title: No Sedation Versus Daily Interruption of Sedation in Chronic Obstructive Pulmonary Disease Mechanically Ventilated Patients- A Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Abeer Abdulghani Soliman Mohammed Emara, assistant lecturer, Benha University
Other Study IDs: MD 9-11-2024
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Sedation and Analgesia
Keywords: Choronic Obstructive Pulmonary disease (COPD); sedation and analgesia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- The patients will be managed by DIS. Richmond agitation and sedation score (RASS) will be used for m: This group of patients will be managed with the no sedation protocol. If agitation occurred, searching for a cause of patient discomfort will be carried out (e.g., tube obstruction or migration, hypoxia, and pain), and managed accordingly. The patient will be reassured and allowed to see his relatives for psychological support if needed, and physical restraints will never be used. If the patient remained agitated, he/she receive IV a bolus of midazolam of 0.5-5 mg as needed to get comfortable and calm. Afterwards, we will start a new trial of management with no sedation; if the sedation has to be repeated three times, we will keep the patient sedated by DIS protocol according to the control group protocol. We will not allow crossover between the groups. We will keep the shifted patients to the DIS protocol after failure of no-sedation protocol in their parent group according to the intention to treat principle.
  Interventions: Behavioral: daily Interruption of Sedation

INTERVENTIONS:
Behavioral: daily Interruption of Sedation — The patients will be managed by DIS. Richmond agitation and sedation score (RASS) will be used for monitoring the depth of sedation

SUMMARY:
this study is to compare no-sedation versus daily interruption of sedation (DIS) in Chronic obstructive pulmonary disease (COPD) patients receiving mechanical ventilation upon the ventilator-free days.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sex aged 18 years or older
* The study will include 60 patients divided into 2 equal groups
* Invasive mechanical ventilation
* Patients with COPD patients (post-bronchodilator FEV1/FVC< 70, and under follow through the department outpatient clinic) exacerbation admitted to the ICU and required invasive mechanical ventilation were recruited.

Exclusion Criteria:

Allergy to sedative which will be used

* renal or hepatic impairment
* proven or suspected psychiatric or neurological impairment
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 60 patients divided into 2 equal groups
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free days | from day-1 to day-28)
  Ventilator-free days (Number of days from day-1 to day-28) on which the patient did not need assistance to his breathe.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospitals, Banhā, Qalyubia Governorate, Egypt